CLINICAL TRIAL: NCT00875329
Title: TBI Screening Instruments and Processes for Clinical Follow-Up
Brief Title: Traumatic Brain Injury (TBI) Screening Instruments
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SDR 08-411
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Brain Injury
Keywords: Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — As there are no biospecimans, there is no biospeciman description.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: A convenience sample of 97VHA patients who served during the OEF or OIF era, who are targeted in CPRS as requiring the TBI Clinical reminder will be included. This includes all ages, both sexes, and all races and ethnicities.

SUMMARY:
Goal: The ultimate goal of this research program is to improve the health and quality of life for wounded warriors from Operations Enduring Freedom and Iraqi Freedom (OEF/OIF) through screening, risk assessment, and outcome measurement.

Purpose: The purpose of this study is to evaluate the reliability and validity of the existing Traumatic Brain Injury (TBI) Clinical Reminder Screen for OEF/OIF Veterans.

DETAILED DESCRIPTION:
Objectives: To meet a VA-wide need for early diagnosis of mild traumatic brain injuries (TBI) in returning soldiers, in April 2007 VA established policy and procedures for screening and evaluation of possible TBI in OEF and OIF veterans. Although the screening process has been in effect for over a year, the validity, reliability, false positive rates, and false negative rates of the TBI Clinical Reminder are unknown. The purpose of this research is to develop a gold standard and then assess the validity/reliability of the TBI Clinical Reminder screen. Specific short-term objectives for this study include:

1. Operationalize a gold standard for TBI identification, using a national panel of experts.
2. Identify patient characteristics and levels of Polytrauma care that predict a delay in or failure to complete the TBI Clinical Reminder screen
3. Using the gold standard, evaluate the validity (sensitivity and specificity) and reliability of the current TBI Clinical Reminder Screen.
4. Identify approaches to improve the TBI Clinical Reminder screening protocol, including screening instrument and process.

Research Design: Methodologies for this study include both prospective and retrospective approaches. Experts will convene in Tampa to operationalize a gold standard for TBI identification (Objective 1). Retrospective, population-based cohort analyses of extant databases will provide insight into current practices and findings to address Objective 2. The gold standard developed in Objective1 will be implemented with a small time-limited prospective cohort so that psychometric analysis of the TBI screen can be conducted (Objective 3). Findings from these analyses will help identify potential improvement in the TBI Screening process to address Objective 4.

Collaboration: This study is responsive to the RFP (#410127, TBI Screen, 8/7/2008). The Tampa HSR&D REAP is partnering with investigators at the Boston VAMC; Tampa investigators are taking the lead on the psychometric evaluation of the TBI screen, while Boston investigators will use the same cohort to evaluate the Second Level TBI Evaluation. Researchers from both sites are co-investigators on each of the proposals to enhance collaboration and linkage of findings.

Anticipated Impact: Traumatic brain injury (TBI), and particularly mild TBI, is said to be the "signature injury" of the current conflicts. These injuries are currently a focus of post-deployment assessment and treatment within the VA and are likely to continue to be the focus of treatment for many years to come. To ensure that OEF/OIF veterans with TBI are identified and treated, the VA TBI Clinical Reminder was instituted in the form of a four-item screening tool for use in VA. While the VA-TBI screening reminder rolled out on April 2, 2007, the utility and psychometric properties of this screening are unknown. The proposed project will address these gaps by operationalizing a gold standard for TBI identification and then using that gold standard to evaluate the reliability and validity of the current TBI screen. By completing this project, we propose to identify specific improvements to the TBI protocol instrument and screening process.

ELIGIBILITY:
Inclusion Criteria:

* Served in OEF/OIF

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All those who have served in OEF/OIF who have been or need to be screened using the TBI Clinical Reminder
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney D. Vanderploeg, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

REFERENCES:
- [Result] Belanger HG, Vanderploeg RD, Soble JR, Richardson M, Groer S. Validity of the Veterans Health Administration's traumatic brain injury screen. Arch Phys Med Rehabil. 2012 Jul;93(7):1234-9. doi: 10.1016/j.apmr.2012.03.003. Epub 2012 Mar 15. PMID 22426242
- [Result] Vanderploeg RD, Groer S, Belanger HG. Initial developmental process of a VA semistructured clinical interview for TBI identification. J Rehabil Res Dev. 2012;49(4):545-56. doi: 10.1682/jrrd.2011.04.0069. PMID 22773258

RESULTS

PARTICIPANT FLOW:
Groups:
- Convenience Sample: A convenience sample of 97VHA patients who served during the OEF or OIF era, who are targeted in CPRS as requiring the TBI Clinical reminder were included. This included all ages, both sexes, and all races and ethnicities. All participants provided responses to demographic information, a TBI Re-screen, and a semi-structured TBI Identification Clinical Interview.
Period: Overall Study
Arm/Group | Convenience Sample
Started | 97
Completed | 97
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 87

OUTCOME MEASURES:

1. Primary Outcome: Responses From the TBI Clinical Reminder
Description: The presence or absence of symptomatic TBI as determined by the VA TBI Clinical Reminder screen was compared to presence or absence of a deployment-related TBI as determined by the study's criterion standard (i.e., the VA TBI Clinical Identification Interview) to determine concordance and calculate sensitivity and specificity of the VA TBI Clinical Reminder screen. Sensitivity of the screen was the percent of positive screens of those determined to be true positives by the VA TBI Clinical Identification Interview. Specificity was the percentage of negatives screens that were determined to be true negatives by the VA TBI Clinical Identification Interview.
Time Frame: April 2007 January 2012
Measure: Number; unit: percentage of participants
Groups:
- Convenience Sample: A convenience sample of 97VHA patients who served during the OEF or OIF era, who are targeted in CPRS as requiring the TBI Clinical reminder will be included. This includes all ages, both sexes, and all races and ethnicities.
Arm/Group | Convenience Sample
Number analyzed (Participants) | 97
percentage of participants
  Sensitivity | 61
  Specificity | 88

ADVERSE EVENTS:
Time Frame: Overall study: April 2007 to present
Description: Data collection was paper-and-pencil demographic and TBI Screening followed by a semi-structured TBI Identification Clinical Interview.
Groups:
- Convenience Sample: A convenience sample of 97 VHA patients who served during the OEF or OIF era, who are targeted in CPRS as requiring the TBI Clinical reminder will be included. This includes all ages, both sexes, and all races and ethnicities.
Arm/Group | Convenience Sample
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes